CLINICAL TRIAL: NCT07211971
Title: the Value of Flexible Bronchoscopy in the Neonatal Intensive Care Unit at Sohag University Hospitals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hager Khaled Abdelmonem, Resident physician in the Department of Pediatrics and Neonatology, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-25-9-10MS
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Study Including Neonates Who Underwent Flexible Fiberoptic Bronchoscopy in Last 10 Years at Sohag University Hospitals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neonates who underwent flexible fiberoptic bronchoscopy (Other)
  Interventions: Diagnostic Test: retrospective study including neonates who underwent flexible fiberoptic bronchoscopy over a period of 10 years from January 2015 to January 2025.

INTERVENTIONS:
Diagnostic Test: retrospective study including neonates who underwent flexible fiberoptic bronchoscopy over a period of 10 years from January 2015 to January 2025. — retrospective study including neonates who underwent flexible fiberoptic bronchoscopy over a period of 10 years from January 2015 to January 2025.

SUMMARY:
The aim of this study to describe the utility of flexible fiberoptic bronchoscopy for the diagnosis and management of different respiratory diseases in the neonatal ICU.

DETAILED DESCRIPTION:
Study including neonates who underwent flexible fiberoptic bronchoscopy over a period of 10 years from January 2015 to January 2025. The study population comprised neonates admitted to the NICU in Sohag University Hospitals between January 2015 and january 2025.

* The inclusion criteria were neonates aged from 1 day to 28 days with recurrent dyspnea, stridor, recurrent chocking or suspicious respiratory tract anomaly; with recurrent pulmonary infection or atelectasis in the same lung lobe; with suspicious tracheal stenosis in radiological image [X-ray or computed tomography (CT) scan]; inability to be extubated without clear reason; or confirmed congenital esophageal atresia to clarify the presence and position of esophagobronchial fistula before surgery.
* Exclusion criteria : neonates with neurological , cardiac problem ,age above 28 days Clinical data such as age, sex; weight at bronchoscopy; mechanical ventilation during hospitalization.
* Clinical indications and results of bronchoscopy were also retrospectively collected.
* Medical and surgical intervention needed for management after diagnosis by FB.

ELIGIBILITY:
Inclusion Criteria:

* neonates aged from 1 day to 28 days with recurrent dyspnea, stridor, recurrent chocking or suspicious respiratory tract anomaly; with recurrent pulmonary infection or atelectasis in the same lung lobe; with suspicious tracheal stenosis in radiological image [X-ray or computed tomography (CT) scan]; inability to be extubated without clear reason; or confirmed congenital esophageal atresia to clarify the presence and position of esophagobronchial fistula before surgery.

Exclusion Criteria:

neonates with neurological , cardiac problem ,age above 28 days

-

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
the number of patients underwent flexible bronchoscopy in NICU at sohag university hospitals | immediatly after bronchoscopy
  this study conducted to detrmine the number of patient underwent flexible bronchoscopy and importance of flexible bronchoscopy to reach final diagnosis and help in management of different respiratory diseases in NICU at sohag university hospitals by using the documented data including (number of patients, result of bronchoscopy of each patient as diagnosis and treatment)
diagnosis of each neonate which reached by the broncscopy | immediatly after bronchoscopy
  this study conducted to detrmine the number of patient underwent flexible bronchoscopy and importance of flexible bronchoscopy to reach final diagnosis and help in management of different respiratory diseases in NICU at sohag university hospitals by using the documented data including (number of patients, result of bronchoscopy of each patient as diagnosis and treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No